CLINICAL TRIAL: NCT02032160
Title: Study to Generate Exploratory Training Data Characterising Innate/ Adaptive Immune Responses Following 1st & 3rd Intra-muscular Immunisations With Fendrix/Engerix B Vaccines in Healthy Adult Males With no Pre-existing Immunity to Hep B
Brief Title: A Study to Characterise Immune Responses Following Immunisations With "Fendrix" or "Engerix B" Hepatitis B Vaccines
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Surrey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: CRC306B
Record Dates: First submitted 2013-06-18; First posted 2014-01-09 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-02

CONDITIONS: Hepatitis B
Keywords: ADITEC; Immunology; Vaccines; Hepatitis B; Investigational study; innate and adaptive immune responses; Hepatitis B vaccinations
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Engerix B (Experimental): Engerix B IM injection - 20ug At 0, 1 and 6 months
  Interventions: Biological: Engerix B IM injection - 20ug
- Fendrix (Experimental): Fendrix IM injection - 20ug At 0, 1 and 6 months
  Interventions: Biological: Fendrix IM injection - 20ug

INTERVENTIONS:
Biological: Engerix B IM injection - 20ug — Engerix B IM injection - 20ug At 0, 1 and 6 months
  Arms: Engerix B
Biological: Fendrix IM injection - 20ug — Fendrix IM injection - 20ug At 0, 1 and 6 months
  Arms: Fendrix

SUMMARY:
The purpose of this study is to generate an exploratory training set of data and to identify predictive biomarkers (a measurable biological response that predicts something) of innate and adaptive responses to immunisation of two vaccines utilizing different adjuvant technology given according to approved schedules to healthy adult volunteers. The vaccines are model agents selected as they match antigens but have discordant adjuvants, have a known immunogenicity profile, assays are freely available to measure responses, and they are safe to administer to healthy adults at the doses and schedules proposed. This study will strive to correlate biomarker activity with observed immunological responses to vaccination and if successful, these biomarkers could be used in early stage clinical trials to optimize selection of vaccine candidates with a profile that will be most likely to be effective once they are in generalized use.

DETAILED DESCRIPTION:
The purpose of this study is to generate an exploratory training set of data and to identify predictive biomarkers (a measurable biological response that predicts something) of innate and adaptive responses to immunisation of two vaccines utilizing different adjuvant technology given according to approved schedules to healthy adult volunteers. The vaccines are model agents selected as they match antigens but have discordant adjuvants, have a known immunogenicity profile, assays are freely available to measure responses, and they are safe to administer to healthy adults at the doses and schedules proposed. This study will strive to correlate biomarker activity with observed immunological responses to vaccination and if successful, these biomarkers could be used in early stage clinical trials to optimize selection of vaccine candidates with a profile that will be most likely to be effective once they are in generalized use.

In this study, 15 subjects per vaccine will be recruited to receive immunization with one of two hepatitis B vaccines, Engerix B or Fendrix, representing exactly matched antigens (hepatitis B surface antigen) but discordant adjuvant technologies. Following a screening visit, subjects will be randomly allocated to receive three doses of a vaccine at 0, 1 and 2 months. Innate immune responses (cytokine levels and whole blood gene expression) after doses #1 and #3 and adaptive immune responses (serum antibody and antigen specific cellular responses) will be measured at various timepoints after immunisation on an outpatient basis.

The study is funded by ADITEC, which is a collaborative research programme that aims to accelerate the development of novel and powerful immunisation technologies for the next generation of human vaccines.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects aged 18-55 years inclusive
2. The subject is, in the opinion of the investigator, healthy on the basis of a physical examination, medical history, blood results, vital signs, with no active disease process that could interfere with the study endpoints.
3. The subject is able to read and understand the Informed Consent Form (ICF), and understand study procedures.
4. The subject has signed the ICF.
5. The subject has not previously received a vaccine for Hepatitis B or contracted Hepatitis B infection.
6. The subject is seronegative to Hepatitis B as confirmed at screening by assessments of sAb, sAg, and cAb.
7. Seronegative for HIV 1 & 2 antibodies and hepatitis C antibodies at screening.
8. Available for follow-up for the duration of the study.
9. Agree to abstain from donating blood during and for three months after the end of their participation in the study, or longer if necessary.
10. Visa long enough allowing them to complete the study (if applicable).
11. The subject has venous access sufficient to allow blood sampling as per the protocol.

Exclusion Criteria:

1. Known hypersensitivity to any component of the vaccines (excipients: sodium chloride, disodium phosphate dehydrate, sodium dihydrogen phosphate; adjuvants: aluminium phosphate, AS04C, aluminium hydroxide; Hepatitis B antigen produced in yeast cells) or subjects who have exhibited hypersensitivity to any other Hepatitis B vaccine, or a history of any allergy that in the opinion of the investigator would contraindicate subject participation.
2. Presence of primary or acquired immunodeficiency states with a total lymphocyte count less than 1,200 per mm3 or presenting other evidence of lack of cellular immune competence e.g. leukaemias, lymphomas, blood dyscrasias, or patients receiving immunosuppressive therapy (including regular use of oral, inhaled, topical or parenteral corticosteroids).
3. Use of any immune suppressing or immunomodulating drugs within 6 months of Visit 1 (screening).
4. Regular use of non-steroidal anti-inflammatory drugs (by any route of administration including topical) within 6 months of Visit 1 (screening) considered by the study physician as likely to interfere with immune responses.
5. Receipt of a vaccine within 30 days of visit 2. Other vaccines (e.g. for travel) may be administered between visit 13 and 14 only.
6. Currently participating in another clinical study with an investigational or non-investigational drug or device, or has participated in a clinical study within the 3 months preceding Visit 1.
7. Any condition that, in the investigator's opinion, compromises the subject's ability to meet protocol requirements or to complete the study.
8. Receipt of blood products or immunoglobin, or blood donation, within 3 months of screening.
9. Unable to read and speak English to a fluency level adequate for the full comprehension of procedures required in participation and consent.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-05; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Change from pre-immunisation baseline values in global gene expression measured on whole blood samples. | visit 2 - 14 (Day 0, 1, 3, 7, 14, 28, 56, 57, 59, 63, 70, 84 and 168).

SECONDARY OUTCOMES:
Change from pre-immunisation baseline values in serum anti-hepatitis B IgG (immunoglobulin G) titre in serum samples. | visit 2 - 14 (Day 0, 1, 3, 7, 14, 28, 56, 57, 59, 63, 70, 84 and 168).

OTHER OUTCOMES:
Change from pre-immunisation baseline values in metabolic gene expression and pathway activation measured on whole blood samples. | visit 2 - 14 (Day 0, 1, 3, 7, 14, 28, 56, 57, 59, 63, 70, 84 and 168).
Change from pre-immunisation baseline values in concentration of selected cytokines and acute phase proteins in serum samples. | visit 2 - 14 (Day 0, 1, 3, 7, 14, 28, 56, 57, 59, 63, 70, 84 and 168).
Change from pre-immunisation baseline values in PBMC (peripheral blood mononuclear cell) cytokine secretion, proliferation or surface markers in response to in vitro antigen stimulation. | visit 2 - 14 (Day 0, 1, 3, 7, 14, 28, 56, 57, 59, 63, 70, 84 and 168).
Fold increase in serum hepatitis B IgG titre | visit 2 - 14 (Day 0, 1, 3, 7, 14, 28, 56, 57, 59, 63, 70, 84 and 168).
Correlations in changes in innate immune activation with adaptive immune responses | visit 2 - 14 (Day 0, 1, 3, 7, 14, 28, 56, 57, 59, 63, 70, 84 and 168).

CONTACTS AND LOCATIONS:
Overall Officials: David JM Lewis, MD, Principal Investigator — University of Surrey
Locations (1):
- Surrey Clinical Research Centre, Guildford, Surrey, United Kingdom